CLINICAL TRIAL: NCT04016545
Title: Mortality and Complications in Endovascular Procedures Performed With New Generation Low-profile Devices
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Associate Professor of Vascular Surgery, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 30027/19
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Peri-operative Mortality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treated patients
  Interventions: Device: Low profile endoprothesis (Navion Medtronic, NBS Low Profile Bolton Terumo)

INTERVENTIONS:
Device: Low profile endoprothesis (Navion Medtronic, NBS Low Profile Bolton Terumo) — Aortic aneurysm exclusion through endovascular procedure

SUMMARY:
The aim of this study is to observe mortality and complications in procedures in which are used new generation low-profile endoprothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indications for elective TEVAR

Exclusion Criteria:

* Incapability to provide consent
* Patients not eligible for TEVAR
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients eligible for elective TEVAR treatable with low-profile endoprothesis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Post-operative mortality (intra-operatory and up to 30 days post-surgery)

SECONDARY OUTCOMES:
Complications | 24 months
  Complications during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided